CLINICAL TRIAL: NCT02529410
Title: A Multicentre Randomised Control Trial Comparing Standard Cardiac Resynchronisation Pacing With Triventricular Pacing
Brief Title: Standard Care Versus Triventricular Pacing in Heart Failure
Acronym: STRIVE HF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/LO/0183
Record Dates: First submitted 2015-08-17; First posted 2015-08-20 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy; Defibrillators

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triventricular pacing (Experimental): 2 Left ventricular leads and one right ventricular lead
  Interventions: Procedure: Cardiac Resynchronisation Therapy
- Biventricular leads (Active Comparator): 1 left ventricular lead and one right ventricular lead
  Interventions: Procedure: Cardiac Resynchronisation Therapy

INTERVENTIONS:
Procedure: Cardiac Resynchronisation Therapy
  Other Names: Cardiac Resynchronisation Therapy with Defibrillator

SUMMARY:
100 pt multicentre study 50 pts randomised to triventricular pacemaker, 50 to biventricular pacemaker Feasibility study with 6 month outcome data

DETAILED DESCRIPTION:
100 patients with QRS duration (120-150ms LBBB) for device insertion as per ESC guidelines 2013 will be recruited to the study from 10 centres. Patients will undergo the pre-operative work up that is typical of their institution (for example at the GSTT site this will include cardiac MRI, cardiopulmonary exercise testing (CPET), 6 minute walk test , bloods including Nt pro BNP, Minnesota living with heart failure questionnaire (MLWHFQ), 2D/3D echocardiogram and the collection of demographic data.)

Patients will then be randomised in a 1:1 fashion to receive either the Triventricular device or the conventional biventricular device.

Participants will then be followed up as per the implanting institution's typical follow up. (for example at GSTT this will include 6 week atrio-ventricular and ventricular-ventricular optimisation (if patients have a device that does not autooptimise) and review by a clinician as well as a 6 month follow up at which point the CPET, 6 minute walk test , MLWHFQ, bloods including Nt pro BNP, 2D/3D echocardiogram and the collection of demographic data will be repeated.)

Regardless of the institution's own follow up, a 6 week (4-8 week) and 6 month (5-9month) follow up appointment will form part of the study protocol. The 6 week check will be take the form of a standard clinical pacing check with physician input if it is deemed necessary as per the host institution's usual standard of care/ (usually one would imagine if a problem of therapy delivery is noted)

The 6 month follow up will allow for patient and device follow up. This will require 2D echocardiography, 6 min walk test, MLWHFQ and NtproBNP measurement. Where possible institutions will be encouraged to perform CPET and 3D echocardiography pre implant and at 6 months.

For determining the " response rate", a positive response will be defined as an absolute reduction of LVESV by 15%. In order to determine the magnitude of response then the change in LVESV will be assessed as a continuous variable.

ELIGIBILITY:
Inclusion Criteria:

* Class 1b Indication for CRT (LBBB QRS120-150ms) as per ESC guidelines 2013
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Insufficient capacity to consent to the study
* QRS >150ms and Non-LBBB morphology 120-150ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of achieving and maintaining triventricular pacing at 6 months | 6 months
  Percentage of patients having triventricular pacing at 6 months

SECONDARY OUTCOMES:
Proportion of patients who successfully reverse remodel as per echo (success being defined as a reduction in end systolic volume of > 15% | 6 months
  outcome
Proportionate effect of intervention and comparator with regard to reverse remodelling (comparison of % reduction in left ventricular end systolic volume ) | 6 months
  outcome
Proportion of patients who successfully reverse remodel as per echo (success being defined as a reduction in end systolic volume of > 15% with prespecified subgroups (AF and aetiology) | 6 months
  6 months
Proportionate effect of intervention and comparator with regard to reverse remodelling (comparison of % reduction in left ventricular end systolic volume ) (AF and aetiology) | 6 months
  outcome
Mean change in Nt proBNP in patients with triventricular devices compared with biventricular devices (pg/ml) | 6 months
  outcome
Comparison of effect of biventricular and triventricular pacing on scores in the Minnesota Living with Heart Failure Questionnaire | 6 months
  outcome
Comparison of effect of biventricular and triventricular pacing on change in 6 minute walk test (metres) | 6 months
  outcome
Percentage change in Nt proBNP in patients with triventricular devices compared with biventricular devices | 6 months
  outcome
Comparison of percentage of shocks delivered in triventricular arm vs biventricular arm | 6 months
  outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas Hospital Trust, London, United Kingdom

REFERENCES:
- [Derived] Gould J, Claridge S, Jackson T, Sieniewicz BJ, Sidhu BS, Porter B, Elliott MK, Mehta V, Niederer S, Chadwick H, Kamdar R, Adhya S, Patel N, Hamid S, Rogers D, Nicolson W, Chan CF, Whinnett Z, Murgatroyd F, Lambiase PD, Rinaldi CA. Standard care vs. TRIVEntricular pacing in Heart Failure (STRIVE HF): a prospective multicentre randomized controlled trial of triventricular pacing vs. conventional biventricular pacing in patients with heart failure and intermediate QRS left bundle branch block. Europace. 2022 May 3;24(5):796-806. doi: 10.1093/europace/euab267. PMID 35079787